CLINICAL TRIAL: NCT04076683
Title: Validation d'Une Stratégie de Programme Transfusionnel Par Erythraphérèse basée Sur un Algorithme d'Aide à la Prescription Transfusionnelle Chez Les Patients Adultes Drépanocytaires
Brief Title: Algorithm for Apherisis Monitoring and Prescription Assistance in Sickle Cell Patients (ALGODREP)
Acronym: ALGODREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etablissement Français du Sang (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Paris 12 Val de Marne University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-A01411-50
Record Dates: First submitted 2019-08-26; First posted 2019-09-03 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Sickle Cell Disease
Keywords: Algorithm; Apherisis; Sickle cell patients
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algorithm (arm A) (Experimental): Frequency and volume for apherisis proposed by algorithm and validated by the physician
  Interventions: Device: Algodrep
- Usual care (arm C) (No Intervention): Frequency and volume for apherisis only decided by the physician (usual care)

INTERVENTIONS:
Device: Algodrep — Algorithm computing the volume of blood to be transfused and the interval between apheresis which are necessary to maintain an individual objective of HbS percentage.
  Arms: Algorithm (arm A)

SUMMARY:
The main objective of this study is to prove the superiority of a procedure which calculates the volume of RBCs to transfuse and the time between apheresis based on this algorithm, compared to the current procedure. The primary endpoint would be the number of patients with individually achieved objectives in terms of % HbS before each apheresis (which reflects the effectiveness of the previous apheresis) over a period of 12 months. The secondary objectives would be to compare the volume differences of transfused RBCs in both groups over a period of 12 months, the occurrence of clinical events and the satisfaction of patients and physicians.

The investigators hope that this study would improve the efficiency and the performance of apheresis in sickle cell patients. The investigators also hope to facilitate the organization of procedures with the flexibility that would allow the use of this algorithm.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is the most common genetic disease leading to abnormal hemoglobin (HbS). Chronic complications can be severe and affect multiple organs. Among them, cerebrovascular disease is one of the most serious leading to a high risk of stroke. These complications often require blood exchange transfusions (BET) in order to replace red blood cells (RBC) containing HbS (from patients) by GR containing HbA (blood donors), and thereby stop the harmful pathophysiological cascade. The indications of long-term apheresis are mostly, but not exclusively, represented by cerebral vasculopathy (85% in our center), and chronic organ damages. Long-term BET in cerebral vasculopathy may considerably reduce the risk of stroke while stopping them leads to a recurrence of this risk, hence there is a need to do them regularly (on average every 4 to 6 weeks) with an objective of HbS ≤ 30%. This objective may be less stringent in the case of other indications.

Two methods are used: a manual method which is feasible anywhere and the apheresis which is preferred because of its better efficacy in achieving the targets of HbS percentage. It also limits transfusion hemochromatosis.

The volume required for BET by apheresis as well as the optimal period between apheresis sessions are empirically determined.

In our practice, the investigators noticed that this method did not allow to steadily obtaining the %HbS objective and the interval between apheresis was variable, in part conditioned by the availability of machines. This implies a real risk of occurrence of recurrent stroke in patients with cerebral vascular disease and may cause a lack of flexibility in the timing of appointments.

Thereby the principal investigator and the biostatistician created an algorithm to compute the volume of blood to be transfused and the interval between apheresis which are necessary to maintain an individual objective of HbS percentage. This algorithm has been obtained by statistical analysis of apheresis performed at Henri Mondor Hospital over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have sickle cell disease, defined as those individuals with HbSS or HbSβ0Thal
* Included in a Blood Exchange Transfusion program (apherisis)
* Benefiting from social insurance
* Accepting to participate in the study and having signed the informed consent

Exclusion Criteria:

* Have sickle cell disease defined with S-β+thal
* Receiving EPO treatment
* Pregnant or breast-feeding women
* Lack of effective contraception in women in childbearing age
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with individually achieved objectives in terms of % HbS | For each apherisis over a 12 months period

SECONDARY OUTCOMES:
Volume of transfused RBCs | For each apherisis over a 12 months period
Number of transfused RBCs | For each apherisis over a 12 months period
Number of apherisis per participant | Over a 12 months period
Hematocrit (percentage) | For each apherisis over a 12 months period
Hemoglobin (g/dL) | For each apherisis over a 12 months period
Number of reticulocyte (g/L), | For each apherisis over a 12 months period
Percentage of reticulocyte | For each apherisis over a 12 months period
Lactate dehydrogenase (UI/L) | For each apherisis over a 12 months period
Creatinine (mg/L) | For each apherisis over a 12 months period
Alanine aminotransferase (UI/L) | For each apherisis over a 12 months period
Aspartate aminotransferase (UI/L) | For each apherisis over a 12 months period
Bilirubin T (mg/dL) | For each apherisis over a 12 months period
Percentage of alloimmunisation events evaluated with irregular red cell antibodies measure | For each apherisis over a 12 months period
Quality of life questionnaire (SF-36) | At baseline and in 12 months
Physician satisfaction survey for each participant | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Pablo BARTOLUCCI, Principal Investigator — Henri Mondor University Hospital
Locations (8):
- France (7):
  - EFS Rhône-Alpes-Auvergne, Saint-Priest-en-Jarez, Auvergne-Rhône-Alpes
  - Centre de Santé EFS, Besançon, Bourgogne-Franche-Comté
  - Centre de Santé EFS, Rennes, Brittany Region
  - Centre de Santé EFS, Tours, Centre-Val de Loire
  - Centre de Santé EFS, Bordeaux, Nouvelle-Aquitaine
  - Hôpital Henri Mondor, Créteil, Île-de-France Region
  - CHU Kremlin Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
- CHU de Martinique, Le Lamentin, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quinn CT, Ahmad N. Clinical correlates of steady-state oxyhaemoglobin desaturation in children who have sickle cell disease. Br J Haematol. 2005 Oct;131(1):129-34. doi: 10.1111/j.1365-2141.2005.05738.x. PMID 16173973
- [Background] Quinn CT, Sargent JW. Daytime steady-state haemoglobin desaturation is a risk factor for overt stroke in children with sickle cell anaemia. Br J Haematol. 2008 Feb;140(3):336-9. doi: 10.1111/j.1365-2141.2007.06927.x. Epub 2007 Nov 27. PMID 18042265
- [Background] Setty BN, Stuart MJ, Dampier C, Brodecki D, Allen JL. Hypoxaemia in sickle cell disease: biomarker modulation and relevance to pathophysiology. Lancet. 2003 Nov 1;362(9394):1450-5. doi: 10.1016/S0140-6736(03)14689-2. PMID 14602439
- [Background] Nahavandi M, Nichols JP, Hassan M, Gandjbakhche A, Kato GJ. Near-infrared spectra absorbance of blood from sickle cell patients and normal individuals. Hematology. 2009 Feb;14(1):46-8. doi: 10.1179/102453309X385133. PMID 19154664
- [Background] Nahavandi M, Tavakkoli F, Hasan SP, Wyche MQ, Castro O. Cerebral oximetry in patients with sickle cell disease. Eur J Clin Invest. 2004 Feb;34(2):143-8. doi: 10.1111/j.1365-2362.2004.01307.x. PMID 14764078
- [Background] Waltz X, Pichon A, Lemonne N, Mougenel D, Lalanne-Mistrih ML, Lamarre Y, Tarer V, Tressieres B, Etienne-Julan M, Hardy-Dessources MD, Hue O, Connes P. Normal muscle oxygen consumption and fatigability in sickle cell patients despite reduced microvascular oxygenation and hemorheological abnormalities. PLoS One. 2012;7(12):e52471. doi: 10.1371/journal.pone.0052471. Epub 2012 Dec 20. PMID 23285055
- [Background] Waltz X, Pichon A, Mougenel D, Lemonne N, Lalanne-Mistrih ML, Sinnapah S, Tarer V, Tressieres B, Lamarre Y, Etienne-Julan M, Hue O, Hardy-Dessources MD, Connes P. Hemorheological alterations, decreased cerebral microvascular oxygenation and cerebral vasomotion compensation in sickle cell patients. Am J Hematol. 2012 Dec;87(12):1070-3. doi: 10.1002/ajh.23318. Epub 2012 Aug 22. PMID 22911571
- [Background] Belcher JD, Chen C, Nguyen J, Milbauer L, Abdulla F, Alayash AI, Smith A, Nath KA, Hebbel RP, Vercellotti GM. Heme triggers TLR4 signaling leading to endothelial cell activation and vaso-occlusion in murine sickle cell disease. Blood. 2014 Jan 16;123(3):377-90. doi: 10.1182/blood-2013-04-495887. Epub 2013 Nov 25. PMID 24277079
- [Background] Eltzschig HK, Carmeliet P. Hypoxia and inflammation. N Engl J Med. 2011 Feb 17;364(7):656-65. doi: 10.1056/NEJMra0910283. No abstract available. PMID 21323543
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429
- [Background] Lionnet F, Arlet JB, Bartolucci P, Habibi A, Ribeil JA, Stankovic K; groupe de recommandations et d'etude de la drepanocytose de l'adulte (GREDA). [Guidelines for management of adult sickle cell disease]. Rev Med Interne. 2009 Sep;30 Suppl 3:S162-223. doi: 10.1016/j.revmed.2009.07.001. Epub 2009 Aug 26. French. PMID 19713011
- [Background] Adams RJ, McKie VC, Hsu L, Files B, Vichinsky E, Pegelow C, Abboud M, Gallagher D, Kutlar A, Nichols FT, Bonds DR, Brambilla D. Prevention of a first stroke by transfusions in children with sickle cell anemia and abnormal results on transcranial Doppler ultrasonography. N Engl J Med. 1998 Jul 2;339(1):5-11. doi: 10.1056/NEJM199807023390102. PMID 9647873
- [Background] Adams RJ, Brambilla D; Optimizing Primary Stroke Prevention in Sickle Cell Anemia (STOP 2) Trial Investigators. Discontinuing prophylactic transfusions used to prevent stroke in sickle cell disease. N Engl J Med. 2005 Dec 29;353(26):2769-78. doi: 10.1056/NEJMoa050460. PMID 16382063
- [Background] Abboud MR, Yim E, Musallam KM, Adams RJ; STOP II Study Investigators. Discontinuing prophylactic transfusions increases the risk of silent brain infarction in children with sickle cell disease: data from STOP II. Blood. 2011 Jul 28;118(4):894-8. doi: 10.1182/blood-2010-12-326298. Epub 2011 Jun 1. PMID 21633086
- [Background] Gueguen A, Mahevas M, Nzouakou R, Hosseini H, Habibi A, Bachir D, Brugiere P, Lionnet F, Ribei JA, Godeau B, Girot R, Ibrahima V, Calvet D, Galacteros F, Bartolucci P. Sickle-cell disease stroke throughout life: a retrospective study in an adult referral center. Am J Hematol. 2014 Mar;89(3):267-72. doi: 10.1002/ajh.23625. PMID 24779035